CLINICAL TRIAL: NCT06740942
Title: Imaging and Serological Biomarkers of Autonomic Dysfunction After Ischemic Stroke
Acronym: ARIADNE
Status: Not yet recruiting | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Eckhard Schlemm, Principal Investigator, Universitätsklinikum Hamburg-Eppendorf
Other Study IDs: 118914145
Record Dates: First submitted 2024-12-14; First posted 2024-12-18 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Acute Ischemic Stroke; Transient Ischemic Attack
Keywords: Autonomic dysfunction; cardiovascular dysregulation; brain-heart axis; stroke-heart syndrome; acute ischemic stroke; transient ischemic attack; autonomic function test; central autonomic network; network lesion mapping; lesion symptom mapping; resting-state fMRI; functional brain network; structural brain network; diffusion tensor imaging
MeSH Terms: conditions — Ischemic Stroke; Ischemic Attack, Transient; Primary Dysautonomias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to

* to investigate the prevalence and time course of autonomic dysfunction in acute ischemic stroke patients;
* to evaluate the influence of lesion location on autonomic dysfunction;
* to identify patterns of structural and functional brain connectivity within the central autonomic control circuits associated with autonomic dysfunction; and
* to explore causal models of the link between brain lesions; cardiac, immunological and endocrine biomarkers; and dysautonomia.

Researchers will compare patients with acute ischemic stroke to patients with transient ischemic attacks to study the effect of acute ischemic brain lesions.

Participants will

* undergo cardiovascular autonomic function testing;
* receive structural and functional MR imaging;
* provide blood samples for determinaton of serological biomarkers auf dysautonomia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of either

  * acute ischemic stroke with either an ischemic lesion visible on CT/MRI or persistent focal deficits 24 hours after symptom onset, or
  * Transient ischemic attack with transient clinical deficits including motor or speech disturbance and not restricted to isolated vertigo/dizziness, visual disturbance, or sensory disturbance.
* symptom onset within 72h prior to hospital admission,
* a pre-stroke/TIA ability to walk without help from another person (modified Rankin scale score < 4),
* age > 18 years, and
* informed consent by either the patient or a legal representative (including a spouse)

Exclusion Criteria:

* In-hospital stroke,
* contraindications to MR imaging (e.g., claustrophobia, pregnancy, pacemakers, implants),
* known moderate to severe dementia,
* previous structural brain damage (except leukoariosis due to cerebral small vessel disease),
* hemodynamically relevant stenosis of the common or internal carotid artery, or
* left heart failure with estimated left ventricular ejection fraction < 50%,
* concomitant systemic illness that can lead to dysautonomia, such as an active infection, thyroid disease, or neurodegenerative disorder (e.g. PD, MSA).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from the Stroke Unit at the Department of Neurology at University Medical Center Hamburg-Eppendorf
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Autonomic dysfunction | 3-5 days after stroke onset
  Cardiovagal and Adrenergic Scores on the Composite Autonomic Scoring Scale (0-7, higher values indicate greater dysfunction)

SECONDARY OUTCOMES:
Autonomic dysfunction | 90 days after stroke onset
  Cardiovagal and Adrenergic Scores on the Composite Autonomic Scoring Scale (0-7, higher values indicate greater dysfunction)

IPD SHARING:
Plan to Share IPD: Yes
All IPD used in the results publication will be shared.
Supporting Information: Analytic Code
Time Frame: IPD and supporting information will be made available with the results publication, and will remain accessible for a minimum of ten years.
Access Criteria: IPD and supporting information will be publically accessible.